CLINICAL TRIAL: NCT00950573
Title: Is Progression of Arteriosclerosis in ESRD Patients Inhibited by Nocturnal Hemodialysis or Renal Transplantation?
Brief Title: Arterial Calcifications in Nocturnal Hemodialysis and Renal Transplantation Versus Conventional Dialysis
Acronym: NOCTX
Status: Completed | Type: Observational
Sponsor: Dianet Dialysis Centers (Other)
Responsible Party: Sponsor
Other Study IDs: NOCTX
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Kidney Disease
Keywords: cardiovascular disease; endstage renal disease
MeSH Terms: conditions — Kidney Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1x 4,5 ml citrate plasma
  1x 10 ml EDTA plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- hemodialysis: patients treated with conventional hemodialysis
- peritoneal dialysis: patients treated with peritoneal dialysis
- nocturnal hemodialysis: patients treated with frequent nocturnal hemodialysis
- kidney transplantation: patients treated with renal transplantation

SUMMARY:
Objective:

1. To assess whether nocturnal hemodialysis and renal transplantation are associated with less progression of coronary arterial calcification, compared with conventional hemodialysis and peritoneal dialysis;
2. To identify the risk factors for coronary arterial calcification in dialysis and transplant patients, and to assess a possible interaction with treatment modality.

DETAILED DESCRIPTION:
To assess whether nocturnal hemodialysis and renal transplantation are associated with less progression of coronary arterial calcification, compared with conventional hemodialysis and peritoneal dialysis; To identify the risk factors for coronary arterial calcification in dialysis and transplant patients, and to assess a possible interaction with treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* ESRD
* current age > 18 and < 75 yr
* ability to understand the study procedures
* willingness to provide written informed consent

Exclusion Criteria:

* life expectancy < 3 months
* claustrophobia
* allergy to iodinated contrast
* treatment incompliance, i.e. non-adherence to dialysis regimens and drug use
* GFR < 30 ml/min (according to MDRD formula) in renal transplant patients
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ESRD
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2010-01; Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Change in coronary artery calcification score | 3 yrs
  The coronary artery calcification score is measured in Agatston units or cubic millimeters and ranges from zero to theoretically infite. This coronary artery calcicifcation score is a total score for all coronary arteries. A higher score, and thus a higher increase in coronary artery calcification score, therefore represents a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Brigit van Jaarsveld, MD, PHD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Dianet Dialysis Centers, Utrecht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided